CLINICAL TRIAL: NCT06078111
Title: Neglect Treatment by Prism Adaptation in the Acute Phase
Acronym: aPA-NEGLECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Roberta Ronchi, Principal Investigator, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: aPA-NEGLECT
Record Dates: First submitted 2023-06-27; First posted 2023-10-11 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Unilateral Spatial Neglect

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prism 10 (Experimental): participants perform rehabilitation activities while wearing 10° visual field deviation prismatic goggles
  Interventions: Behavioral: Prism 10 + visuo-motor activities
- Neutral Prism (Active Comparator): participants perform rehabilitation activities while wearing neutral (no deviation) visual field deviation prismatic goggles
  Interventions: Behavioral: Neutral Prism + visuo-motor activities

INTERVENTIONS:
Behavioral: Prism 10 + visuo-motor activities — Visuo-motor activities of exploration in the left and right space, adapting activities of daily living, while wearing prisms with 10 degrees of visual field deviation
  Arms: Prism 10
Behavioral: Neutral Prism + visuo-motor activities — Visuo-motor activities of exploration in the left and right space, adapting activities of daily living, while wearing prisms with no visual field deviation
  Arms: Neutral Prism

SUMMARY:
This project aims at unveiling the beneficial effects of prism adaptation as early rehabilitation technique to treat unilateral spatial neglect in the acute phase after a brain damage. This syndrome, frequent and very invalidating for daily life activities after a brain damage, is a cognitive disorder of lack of attention towards a part of the space. Patients at a first event brain injury hospitalized into the Neurology and Neurosurgery Departments and affected by spatial neglect will undergo to a protocol of five consecutive rehabilitation treatments, being assigned to the experimental (prisms) or control groups (neutral prisms). The effectiveness of the treatment will be assessed with cognitive, functional and motor-related measures, as well as a follow up 3 months later. These results can have a strong impact on the long-term functional outcome of these patients.

ELIGIBILITY:
Inclusion Criteria:

* First neurological event, affecting the right hemisphere or the left hemisphere (stroke, brain tumour post-surgery);
* Structural images of the brain lesion available (magnetic resonance or tomographic scans);
* Good Normal (or corrected) visual acuity;
* Presence of USN, as assessed by a standard neuropsychological evaluation.

Exclusion Criteria:

* Previous neurological disorder and/or current or previous psychiatric disease.
* Presence or suspicion of previous general cognitive deficits documented from the clinical dossier and/or suspicious of possible cognitive deficits ;
* Presence of difficulty in task's comprehension preventing its completion;
* Impossibility to sustain a research session of at least 30 minutes (e.g., attentional lability).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Unilateral spatial neglect | Day 0; Day 5; 12 weeks after the end of the protocol
  Scores in the neuropsychological tasks administered just before and after the rehabilitation protocol: BEN battery, with the number of lateralized omissions in target cancellation, drawing and reading; bisection bias for the line bisection test
Functional measures | Day 0; Day 5; 12 weeks after the end of the protocol
  Scores in the functional test testing USN administered just before and after the rehabilitation protocol: CBS scale, evaluating the impact of neglect in 10 daily living activities (range 0-30)
Disability measures | Day 0; Day 5; 12 weeks after the end of the protocol
  Scale for assessing disability after stroke just before and after the rehabilitation protocol: FIM (range 18-126)
Balance | Day 0; Day 5; 12 weeks after the end of the protocol
  Balance tests after stroke just before and after the rehabilitation protocol: PASS (range 0-36)

SECONDARY OUTCOMES:
Neuropsychological tests: Right vs. Left neglect | Day 5; 12 weeks after the end of the protocol
  Comparison of the improvements in neuropsychological tests of patients with right vs. left unilateral spatial neglect on the following measures:
  - BEN test: numbers of the lateralized omissions left-right in the target cancellation, drawing, reading; bisection bias in the bisection test The difference between patients with right vs. left spatial neglect following brain damaged will be computed by a difference in the outcome scores (omissions rates, bisection biases) and the incidence (percentage of patients) still defective vs. non-defective at each of these measures
Functional Measures: Right vs. Left neglect | Day 5; 12 weeks after the end of the protocol
  Comparison of the improvements in the functional activities of daily living of patients with right vs. left unilateral spatial neglect on the following measures:
  - CBS scale. The difference between patients with right vs. left spatial neglect following brain damaged will be computed by a difference in the outcome scores (total score of the functional scale) and the incidence (percentage of patients) still defective vs. non-defective at this measure
Disability Measures: Right vs. Left neglect | Day 5; 12 weeks after the end of the protocol
  Comparison of the improvements of the disability scale of patients with right vs. left unilateral spatial neglect on the following measures:
  - FIM The difference between patients with right vs. left spatial neglect following brain damaged will be computed by a difference in the outcome scores (total score of the scale) and the incidence (percentage of patients) still defective vs. non-defective at this measure
Balance: Right vs. Left neglect | Day 5; 12 weeks after the end of the protocol
  Comparison of the improvements of balance of patients with right vs. left unilateral spatial neglect on the following measures:
  - PASS The difference between patients with right vs. left spatial neglect following brain damaged will be computed by a difference in the outcome scores (total score of the scale) and the incidence (percentage of patients) still defective vs. non-defective at this measure
Functional Measures: Follow-up | 12 weeks after the end of the protocol
  Assessment of the functional benefit of the treatment procedure 3-months after the rehabilitation on the following measure:
  - CBS: difference in the total score The difference between patients with spatial neglect who have been submitted to the prism 10 or the neutral prisms protocol will be compared in the follow up. The difference of the scores at the end of the protocol vs. in the follow-up will be performed for each group, and a differential score (prism 10 end of the protocol - prism 10 follow-up vs. neutral prisms end of the protocol - neutral prisms follow-up) will be also analysed to check for the maintenance of the effect. The differences will be computed using the total outcome scores and the incidence (percentage of patients) still defective vs. non-defective at this measure
Balance: Follow-up | 12 weeks after the end of the protocol
  Assessment of the functional benefit of the treatment procedure 3-months after the rehabilitation on the following measure:
  - PASS: difference in the total score The difference between patients with spatial neglect who have been submitted to the prism 10 or the neutral prisms protocol will be compared in the follow up. The difference of the scores at the end of the protocol vs. in the follow-up will be performed for each group, and a differential score (prism 10 end of the protocol - prism 10 follow-up vs. neutral prisms end of the protocol - neutral prisms follow-up) will be also analysed to check for the maintenance of the effect. The differences will be computed using the total outcome scores and the incidence (percentage of patients) still defective vs. non-defective at this measure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland